#### **Patient Consent Form**



# Assessing the Role of Guides in Enhancing Dental Implant Placement Precision and Patient Outcomes

Running title: Fully guided dental implant placement and primary stability

Alyaa I. Naser<sup>1</sup>, Abdulhameed N. Aldabagh<sup>2</sup>, Saif T. Aldabagh<sup>3</sup>

- 1. BDS, MSc. Ph.D., assist. Prof. Department of OMFS, College of Dentistry, University of Mosul, Nineveh, Iraq. <a href="mailto:alyaaismael@uomosul.edu.iq">alyaaismael@uomosul.edu.iq</a>, ORCID: 0000-0001-7051-6836.
- 2. BDS, MSc. Ph.D., assist. Prof. Department of OMFS, College of Dentistry, University of Mosul, Nineveh, Iraq, <a href="mailto:aldaagh@uomosul.edu.iq">aldabagh@uomosul.edu.iq</a> ORCID: 0000-0001-7130-1474.
- 3. BDS, MSc. FIBMS. Lecturer. Department of OMFS, College of Dentistry, University of Mosul, Nineveh, Iraq. Saif tawfik@uomosul.edu.iq, ORCID:0000-0002-9362-6963.

**Funding: self-funding** 

Conflict of interest: no conflict of interest

REC. reference no. UoM. dent. 25/1029

This study was approved by the local ethical committee [Approval letter No. UOM.Dent/25/1029] at 9/12/2024.

University of Mosul College of Dentistry Oral and Maxillofacial Surgery Implant Dental Unit and Laser

#### **Patient Consent Form**



#### Research Ethics Committee



Ministry of Higher Education and Scientific Research University of Mosul College of Dentistry

Date: 09/12/2024

#### **Confirmation Review Letter**

| REC reference no. | UoM.Dent. 25/1029 |
|---|---|
| Project title | Assessing the Role of 3D-Printed Surgical Guides in<br>Enhancing Dental Implant Placement Precision and<br>Patient Outcomes |
| Name of Chief investigator (CI) | Alyaa Ismael Naser |
| Name of principle investigator (PI) | |
| Decision | ☐ Approved. ☐ Pending with request for more information. ☐ Rejected. |
| Validity end date | 1/11/2025 |

#### Dear Applicant,

On behalf of Research Ethics Committee, I can confirm that the committee has reviewed the above project and a permission to commence has been granted on the basis described in the application form as well as on the understanding that the study is conducted in accordance with the research guidelines followed in the university of Mosul/College of Dentistry.

Please note that the approval is considered valid from the date of issuing this letter until the end date specified in the application form. If it is proposed to extend the duration of the study or make a considerable change to the protocol, an amendment notification should be sent to the Committee in advance.

Yours sincerely

9.12.2024

Research Ethics Committee Confirmation Review Letter | Version 1.0 | 1 December 2019

#### **Patient Consent Form**



#### Title of the Study:

.....Assessing the Role of Guides in Enhancing Dental Implant Placement Precision and Patient Outcomes......

#### **Patient Information Sheet**

You are being invited to participate in a clinical research study involving guided dental implant placement using surgical guide technology. This research aims to evaluate the accuracy, healing response, and clinical outcomes of implants placed with computer-generated surgical guides.

## Please read the following information carefully before giving your consent

#### **Purpose of the Study**

This study is being conducted to evaluate the clinical effectiveness and precision of implants placed using surgical guides based on CBCT imaging and digital planning software (e.g., RealGUIDE).

#### **Potential Benefits and Risks**

Benefits: More accurate implant placement, reduced surgical time, and minimal post-operative discomfort.

<u>Risks</u>: As with any surgical procedure, there may be risks of infection, pain, or implant failure. These will be minimized with standard protocols and follow-up.

## Voluntary Participation

Your participation is entirely voluntary. You may choose to withdraw from the study at any time without affecting the quality of your treatment.

## Confidentiality

All your personal information and medical data will be kept strictly confidential and used solely for research purposes.

University of Mosul College of Dentistry Oral and Maxillofacial Surgery Implant Dental Unit and Laser

### **Patient Consent Form**



#### **Declaration and Consent**

I hereby confirm that:

- I have read and understood the information provided above.
- I have had the opportunity to ask questions and receive satisfactory answers.
- I voluntarily agree to participate in this study.
- I understand that I may withdraw at any time without any negative consequences to my care.

| Patient Name: | |
|-------------------------------------|-------|
| Signature: | Date: |
| Researcher/Investigator Name: | |
| Signature: | Date: |
| Ethical Approval | |
| Ethical Committee Approval Stamp | |
| Scientific Committee Approval Stamp | |